CLINICAL TRIAL: NCT04377100
Title: Impact on Anxiety and Motivation of COVID-19 and Predictors of Individual Responses.
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999920112; 20-M-N112
Record Dates: First submitted 2020-05-05; First posted 2020-05-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Anxiety; Healthy Volunteers
Keywords: Coronavirus; Pandemic; Environmental Stress; Avoidance; Healthy Volunteers
MeSH Terms: conditions — Anxiety Disorders; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults 18 and over: Adults 18 and over
  Interventions: Behavioral: Computer task questionnaires

INTERVENTIONS:
Behavioral: Computer task questionnaires — MH COVID-19 Adult, MASQ-SF, STAI, ACS, Hollingshead, DSM XC, PMHC, AUDIT, debriefing questionnaire, and finger-tapping task

SUMMARY:
Background:

Researchers think that people s mental health and behavior will be very affected by the steps taken to slow the spread of COVID-19, such as social distancing. Also, the threat of disease and death, to people and their loved ones, can cause much stress. Researchers want to learn more about these stressors and how they are affecting people.

Objective:

To study the relationship of affective, cognitive, and behavioral responses to stressors related to COVID-19 with neuroimaging and behavioral data collected before COVID-19.

Eligibility:

English-speaking adults age 18 and older

Design:

This online study will include both new participants and those who have taken part in past National Institute of Mental Health studies. All will complete the same surveys and tasks.

Participants will give their name and email address. They will get a username and password. The file that links their username to their personal data will be kept secure.

Participants will complete a set of surveys about the following:

* Sociodemographic data, such age, race, and income
* Education and work status
* Mental and medical illness and treatment
* Family medical history
* Mood
* COVID-19 experience
* Anxiety
* Substance and alcohol use
* Attention control
* Other mental health related topics.

Participants will complete a finger-tapping task. For this, they will press a key a certain number of times in a limited period. They will get to practice the task. After the task, they will complete a survey about it.

It will take about 1 hour to complete the surveys and the task.

About 8 months later, participants will be contacted to repeat the surveys and task.

Compensation is provided.

DETAILED DESCRIPTION:
Study Description:

This protocol has 2 goals: (1) Collect data from NIMH research volunteers who already participated in SNFA neuroimaging studies (protocol 02-M-0321,and 14-M-0114) and examine how individual affective, cognitive, and behavioral responses to COVID-19 can be predicted by neural and clinical measures obtained prior to the pandemic. This part-1 concerns only a limited number of adults and represents a unique opportunity to probe critical questions which are difficult to query in empirical experiments or with only retrospective information on stress experience. (2) Collect a large dataset to examine the impact of COVID-19 stressors on motivation pattern (approach/avoidance behavior) in function of anxiety, cognitive and behavioral responses to the pandemic. This part-2 of the protocol is open to any individuals interested in participating. Overall, this is a time-sensitive research on the impact of environmental stressors generated by the COVID-19 pandemic on anxiety, motivation and potential neural mechanisms informed by predictors. Measures collected consist of ratings of stressors related to COVID-19 and more generally, anxiety, cognition, and behavior, including the performance of a motivation-based task (finger-pressing task). and an attention bias task (dot-probe task). This research will use a study website to consent, survey participants online, and tasks.

Objectives:

The primary objective is to examine the relationship of affective, cognitive and behavioral responses to stressors related to COVID-19 with neuroimaging and behavioral data collected previously, before COVID-19. This research will identify risk and resilience factors (neural and behavioral) among study participants regarding their responses to COVID-19 crisis. The secondary objective is to gather a large dataset to provide information on how sustained environmental stress affect motivated behavior, particularly with respect to biasing behavior towards avoidance, and how individual factors such as anxiety and cognitive function influence the impact on patterns of motivation. These data are expected to help the interpretation of the role of neuroimaging findings.

Endpoints:

The endpoints are 2-fold: anxiety and motivation pattern responses to COVID-19 stressors (1) in function of clinical phenotype; and (2) in function of endophenotype previously collected using high-resolution 7T fMRI. These endpoints will be measured twice using the same online platform approximately 14-20 months after the start of enrollment.

Study Population:

The sample size will be up to 6000 healthy volunteers and anxiety participants. Participants will be males and females, 18 years and older. They must be English-speaking. The study population will include patient and volunteer participants who have consented for an SFNA study in the past (protocols 01-M-0185, 02-M-0321, 03-M-0093 and 14-M-0114), or NIMH healthy volunteer study (17-M-0181) as well as new participants from the general population who respond to advertisements for the SNFA -COVID study but who have not previously been a NIMH study participant. The SNFA -COVID study study participants may or may not be local to the Metropolitan Washington DC area but since the study will be conducted entirely online, this is not relevant.

Description of Sites/Facilities Enrolling Participants:

The protocol is situated at the NIH Clinical Center with no additional supporting sites. The study itself will be conducted entirely online through a secure study website where consent and study measures will be completed and repeated as specified.

Description of Study Intervention:

There are no study interventions as this is a descriptive behavioral health survey study, including questionnaires and computer tasks.

Study Duration:

The estimated time from study initiation to study completion approximately three years.

Participant Duration:

It is expected that participants will participate in the study for up to 14-20 months with an option to recontact in the future.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. 18 years of age and older.
2. Able to read and write English.
3. Able to provide informed consent online using study website.

EXCLUSION CRITERIA:

There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of adult subjects in the U.S.
Sampling Method: Non-Probability Sample
Enrollment: 2962 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Functional connectivity of canonical networks | Date of subject participation
  To examine patterns of neural circuits connectivity as potential predictors of rating scores of affective, cognitive and behavioral (including task performance) responses to COVID-19 among healthy and clinically anxious participants who already participants in SNFA resting-state connectivity studies.

SECONDARY OUTCOMES:
Questionnaire data | Date of subject participation
  To examine how motivational, affective and cognitive function is impacted by COVID-19, and how these responses are influenced by clinical history among a range of participants from a community sample.

CONTACTS AND LOCATIONS:
Overall Officials: Maryland Pao, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We will likely submit the de-identified data to a repository but do not have clear plans yet. We will update as we determine the plans.